CLINICAL TRIAL: NCT03524300
Title: Prospective Randomized Controlled Trial for Comparison of Clinical Efficacy Between Robotic and Laparoscopic Total Gastrectomy in Patients With Clinical Stage I Gastric Cancer
Brief Title: Clinical Efficacy Between Robotic and Laparoscopic Total Gastrectomy in Patients With Clinical Stage I Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of gastric surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-015
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasm; Robotic Surgery
Keywords: Stomach Neoplasm; Robotic Surgery; Total Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Assisted Total Gastrectomy (Experimental): Robotic Assisted Total Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Robotic Assisted Total Gastrectomy
- Laparoscopic Assisted Total Gastrectomy (Active Comparator): Laparoscopic Assisted Total Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic Assisted Total Gastrectomy

INTERVENTIONS:
Procedure: Robotic Assisted Total Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case,robotic assisted total gastrectomy will be performed in the experimental group.
  Arms: Robotic Assisted Total Gastrectomy
Procedure: Laparoscopic Assisted Total Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case,laparoscopic assisted total gastrectomy will be performed in the experimental group.
  Arms: Laparoscopic Assisted Total Gastrectomy

SUMMARY:
The purpose of this study is to explore the clinical efficacy between robotic and laparoscopic total gastrectomy in patients with clinical Stage I gastric cancer

DETAILED DESCRIPTION:
Robotic surgery has been developed with the aim of improving surgical quality and overcoming the limitations of conventional laparoscopy in the performance of complex mini-invasive procedures. The study is designed to explore the clinical outcomes of the robotic assisted total gastrectomy by comparing short- and long-term outcomes including financial cost of robotic and laparoscopic assisted total gastrectomy in the treatment of clinical Stage I gastric adenocarcinoma （cStage IA（T1N0M0）or cStage IB（T1N1M0，T2N0M0））.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy cStage IA（T1N0M0）or cStage IB（T1N1M0，T2N0M0）at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
* The tumor is on the upper or middle third stomach and expected to perform total gastrectomy with D1+/D2-10 lymph node dissction to obtain R0 resection sugicall results.
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) class I to III
* Written informed consent

Exclusion Criteria:

* cStage IIA or more advaned at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* Multiple primary cancer
* History of previous gastric surgery (except ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
* Gastric multiple primary carcinoma
* Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
* History of other malignant disease within the past 5 years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within the past 6 months
* History of cerebrovascular accident within the past 6 months
* History of continuous systematic administration of corticosteroids within 1 month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of the predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  the rate of 3-year disease free survival

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
  the rate of 3-year overall survival rate
3-year recurrence pattern | 36 months
  the pattern of recurrence in 3 years
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
overall postoperative serious morbidity rates | 30 days
  Refers to the incidence of early postoperative complication which is graded as Clavien-Dindo IIIA or higher.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight in kilograms on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory response.
Hospitalization expenses | 30 days
  The cost from admission to discharge
operation time | 1 day
  operation time

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided